CLINICAL TRIAL: NCT06001359
Title: Functional Limitation, Pain, Disability and Quality of Life in Patients With Cervical Spondylotic Radiculopathy
Brief Title: Functional Limitation, Pain and Quality of Life in Patients With Cervical Spondylotic Radiculopathy
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Aydın Sinan Apaydin, Doctor, Karabuk University
Other Study IDs: radiculopathy
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Radiculopathy; Elderly
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Radiculopathy is a neurological condition in which transmission along a spinal nerve and its roots is limited or inhibited. It is most caused by spondylotic changes such as cervical disc herniation leading to nerve root compression, inflammatory changes, and the formation of bony prominences in this region [1]. Pain is the initial symptom and cervical radiculopathy should be suspected when pain radiates from the neck to the shoulder and arm, accompanied by sensory complaints and motor weakness. It is most commonly caused by spondylotic changes, such as cervical disc herniation and bony prominences in this area, leading to nerve root compression and inflammatory changes. Stenotic changes in the spine, which are often observed with aging, can cause nerve damage and compression in individuals, causing radicular pain. However, there is insufficient study in which the relationship between pain caused by cervical spondylotic radiculopathy caused by stenosis and functional disability, disability and quality of life due to radiculopathy in patients is insufficient. In addition, the lack of a comprehensive outcome scale that evaluates the functional limitation caused by radicular pain has also led to a deficiency in the evaluation of functional limitation. In this context, CRES is a newly developed scale used to evaluate functional limitation associated with radicular pain. In this context, in this study, it was aimed to examine the relationship between pain, functional disability, disability and quality of life in patients with cervical spondylotic radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* with lateral-foraminal spinal stenosis in the cervical region
* with or without neck pain consistent with the diagnosis obtained from magnetic resonance imaging
* with unilateral root symptoms such as pain, numbness, weakness in the affected limb, and diagnosis based on MRI and computerized tomography

Exclusion Criteria:

* signs of increased ventral pressure, such as ventral osteophytes, disc calcification, and ligament hypertrophy
* severe neurological deficits, pregnant women, spinal malignancies,
* those who had undergone cervical surgery in the last 12 months
* and those who could not cooperate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 64 patients with spondylotic radiculopathy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Neck/Arm Pain | baseline
  A numeric rating scale will be used to evaluate neck and arm pain severity.
Funcitonal disability | baseline
  The Cervical Radiculopathy Impact Scale (CRIS) will used to determine the functional limitation.
Disability | baseline
  Neck Disability Index (NDI) will used to evaluate the effect of neck pain on activities of daily living
life quality | baseline
  The EuroQol Five-Dimensions - 3-Level (EQ-5D-3L) General Quality of Life Scale will used to evaluate the quality of life of individuals
Severity of stenosis | baseline
  The severity of stenosis will be evaluated with MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Aydın Sinan Apaydın, PhD, Study Director — Assistant Professor
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoomes EJ, Scholten-Peeters GG, de Boer AJ, Olsthoorn RA, Verkerk K, Lin C, Verhagen AP. Lack of uniform diagnostic criteria for cervical radiculopathy in conservative intervention studies: a systematic review. Eur Spine J. 2012 Aug;21(8):1459-70. doi: 10.1007/s00586-012-2297-9. Epub 2012 Apr 25. PMID 22531897
- [Background] Patel EA, Perloff MD. Radicular Pain Syndromes: Cervical, Lumbar, and Spinal Stenosis. Semin Neurol. 2018 Dec;38(6):634-639. doi: 10.1055/s-0038-1673680. Epub 2018 Dec 6. PMID 30522138
- [Background] Kelly JC, Groarke PJ, Butler JS, Poynton AR, O'Byrne JM. The natural history and clinical syndromes of degenerative cervical spondylosis. Adv Orthop. 2012;2012:393642. doi: 10.1155/2012/393642. Epub 2011 Nov 28. PMID 22162812
- [Result] Grasso G, Salli M, Torregrossa F. Does Hybrid Surgery Improve Quality of Life in Multilevel Cervical Degenerative Disk Disease? Five-Year Follow-up Study. World Neurosurg. 2020 Aug;140:527-533. doi: 10.1016/j.wneu.2020.03.097. PMID 32797985
- [Derived] Apaydin AS, Gunes M. Relationships between stenosis severity, functional limitation, pain, and quality of life in patients with cervical spondylotic radiculopathy. Turk J Med Sci. 2024 Jun 6;54(4):727-734. doi: 10.55730/1300-0144.5842. eCollection 2024. PMID 39295627